CLINICAL TRIAL: NCT01269138
Title: Treatment of Congenital Factor VII Deficiency. A Prospective Observational Study
Brief Title: Treatment of Inherited Factor VII Deficiency
Acronym: STER
Status: Completed | Type: Observational
Sponsor: University of L'Aquila (Other)
Collaborators: TRIB s.r.l. (Unknown)
Responsible Party: Principal Investigator, Guglielmo Mariani, Professor of Hematology, University of L'Aquila
Other Study IDs: STERProtocol7.0
Record Dates: First submitted 2010-12-17; First posted 2011-01-04 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Factor VII Deficiency
Keywords: Inherited Factor VII deficiency; Inhibitor development in Factor VII deficiency; Bleeding in Factor VII Deficiency; Surgery in Factor VII deficiency; Prophylaxis in Factor VII Deficiency
MeSH Terms: conditions — Factor VII Deficiency | interventions — Factor VII; recombinant FVIIa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma for Factor VII inhibitor assay is stored and sent to a Central Laboratory for the inhibitor determination. Samples are discharged after the inhibitor determination
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Factor VII Deficient Patients: Patients affected by Inherited Factor VII deficiency undergoing treatment for bleeding episodes, surgery , prophylaxis.Any patient with levels of FVII less than 50% of normal or a mutation known to be associated to a FVII deficiency. Any patient with a FVII deficiency for whom treatment of bleeding episodes, prevention related to surgery and primary/secondary prophylaxis is considered necessary by his/her treating physician can be enrolled.
  Interventions: Drug: plasma derived Factor VII; Drug: recombinant FVIIa; Drug: Fresh Frozen Plasma; Drug: Activated Prothrombin Complex Concentrates; Drug: Virus Inactivated plasma

INTERVENTIONS:
Drug: plasma derived Factor VII — Treatment of bleeding episodes,treatment during surgery and prophylaxis
  Other Names: Facteur VII, LFB (plasma-derived);; Factor VII, PFL (plasma-derived); Factor VII, Baxter Immuno (plasma-derived)
Drug: recombinant FVIIa — Treatment of bleeding episodes,treatment during surgery and prophylaxis
  Other Names: Novoseven
Drug: Fresh Frozen Plasma — Treatment of bleeding episodes,treatment during surgery and prophylaxis
  Other Names: Blood Transfusion Centre Fresh Frozen Plasma
Drug: Activated Prothrombin Complex Concentrates — Treatment of bleeding episodes,treatment during surgery and prophylaxis
Drug: Virus Inactivated plasma — Treatment of bleeding episodes,treatment during surgery and prophylaxis
  Other Names: Octaplas

SUMMARY:
FVII deficiency is a rare coagulation disorder. A limited number of patients are found in most treatment centres and countries. Treatment demands vary considerably amongst FVII deficient patients. Therefore, regular clinical studies will meet with recruitment problems in this particular patient population. The present study intends to elucidate the bleeding patterns in a well-defined collective of FVII deficiency patients who are carefully characterised, to document the actual use of different treatment modalities in different subgroups and to evaluate the efficacy and safety of current available treatment modalities in bleedings, surgery and prophylaxis. The purpose is to gain some evidence based knowledge of treatment of patients with FVII deficiency - an area where treatment decisions are made more on personal clinical experience than on consolidated clinical evidence.

This study intends to register treatment practices as they are actually performed - in a structured and documented way.

DETAILED DESCRIPTION:
To describe the treatment modalities and outcomes of: - bleeding episodes - surgery - prophylaxis in a well defined, international cohort of FVII deficient patients characterised following the methodology used by the International Factor VII deficiency Study Group (IF7SG).

To evaluate the presence (in already treated patients) and/or the appearance of inhibiting antibodies to FVII and/or therapy-related thrombosis.

Study Design:

Prospective observational study on treatment of FVII deficiency patients. This is an outcome study conducted through the procedures set up by the IF7SG, in patients already enrolled or newly enrolled in the database.

Study population and products:

Patients with FVII deficiency (levels of FVII less than 50% of normal or a mutation known to be associated to a FVII deficiency) can be enrolled. All pharmaceutical products considered useful for treatment of FVII deficiency by the centres can be included in the study.

Key assessments:

The database is set up to capture the following assessments, if available:

Bleeding episodes:

• Recording of bleeding location, symptom onset and treatment onset & location • Recording of substitution therapy, concomitant medications and concomitant illness • Recording of 6 hour treatment evaluation for bleeding episodes • Recording of re-bleeding episodes

Surgery/delivery:

• Recording of surgery description , date of surgery and indication • Recording of substitution therapy, concomitant medications and concomitant illness during surgery • Recording of antifibrinolytic drugs used prior, during and/or after surgery •Recording of • Recording of overall treatment evaluation

Prophylaxis:

• Recording of prophylaxis type (primary/secondary), indication for prophylaxis and start/stop date •Recording of prophylaxis therapy, concomitant medications and concomitant illness • Recording of bleeding episodes during prophylaxis •Recording of clinical prophylaxis evaluation

For all:

* Laboratory values (PT/INR, APTT, FVII:C, platelet count, fibrinogen, inhibitor samples) at time points specified in section 7.3.
* Adverse events (including thrombotic events, anaphylactic reactions, DIC reactions, Re- bleedings and mortality)
* Recording of 30 day treatment evaluation (excellent, effective, partly effective, ineffective or not evaluable)
* Duration of hospital stay (ward, ICU) within 30 days after first product treatment • Mortality within 30days after first product administration

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by the patient or next of kin or legally acceptable representative to collect data on treatment of a given bleeding episode, surgical event or prophylactic regimen as specified in the protocol.
* If informed consent is provided by the next of kin or legally acceptable representative, consent must also be obtained from the patient as soon as he/she is able to do so.Informed consent should preferentially be obtained before initiation of treatment or as a minimum before entry of data into the database. 2.Males and females 0 to 90 years of age. 3. Any patient with a FVII deficiency for whom treatment of bleeding episodes, prevention related to surgery and primary/secondary prophylaxis is considered necessary by the treating physician can be enrolled.

Exclusion Criteria:

Ages: 1 Day to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Number of patients affected by inherited Factor VII deficiency to be studied Planned number of patients to be recruited: >200 Planned number of evaluable bleeding episodes >100 Planned number of surgical procedures >50 It is planned to include patients to the registry from all over the world
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2007-01; Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Changes in Factor VII levels | Time 0 (before treatment), 15 minutes and 1 month after treatment
  To describe the treatment modalities and clinical and laboratory outcomes in:
  -bleeding episodes - surgery - prophylaxis in a well defined, international cohort of FVII deficient patients characterised following the methodology used by the IF7SG.

SECONDARY OUTCOMES:
Evaluation of Inhibitor Development | Monthly
  To evaluate the presence (in already treated patients) and/or the appearance of inhibiting antibodies to FVII.

CONTACTS AND LOCATIONS:
Overall Officials: guglielmo mariani, md, Study Director — University of L'Aquila
Locations (1):
- San Salvatore Hospital, L’Aquila, AQ, Italy

REFERENCES:
- [Derived] Morfini M, Batorova A, Mariani G, Auerswald G, Bernardi F, Di Minno G, Dolce A, Fede C, Giansily-Blaizot M, Ingerslev J, Martinowitz U, Napolitano M, Pinotti M, Schved JF; International FVII [IF7] and Seven Treatment Evaluation Registry [STER] Study Groups. Pharmacokinetic properties of recombinant FVIIa in inherited FVII deficiency account for a large volume of distribution at steady state and a prolonged pharmacodynamic effect. Thromb Haemost. 2014 Aug;112(2):424-5. doi: 10.1160/TH13-12-1045. Epub 2014 Apr 24. No abstract available. PMID 24763923
- [Derived] Napolitano M, Giansily-Blaizot M, Dolce A, Schved JF, Auerswald G, Ingerslev J, Bjerre J, Altisent C, Charoenkwan P, Michaels L, Chuansumrit A, Di Minno G, Caliskan U, Mariani G. Prophylaxis in congenital factor VII deficiency: indications, efficacy and safety. Results from the Seven Treatment Evaluation Registry (STER). Haematologica. 2013 Apr;98(4):538-44. doi: 10.3324/haematol.2012.074039. Epub 2013 Feb 12. PMID 23403322